CLINICAL TRIAL: NCT01637896
Title: A Comparison Between Paclitaxel-eluting Balloon in Combination With BMS Implantation vs Conventional Balloon and DES Implantation: the ELICOPTER Trial
Brief Title: A Comparison Between Paclitaxel-eluting Balloon in Combination With BMS Implantation vs Conventional Balloon and DES Implantation
Acronym: ELICOPTER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: the study was halted after an interim analysis perfomed for a perceived excess of target vessel revascularization in the DEB+BMS arm
Sponsor: Leonardo Bolognese, MD (Other)
Responsible Party: Sponsor-Investigator, Leonardo Bolognese, MD, Director, Ospedale San Donato
Organization: Ospedale San Donato (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Arezzo000
Record Dates: First submitted 2012-07-07; First posted 2012-07-11 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DEB+BMS (Experimental): drug-eluting balloon predilation and bare metal stent implantation
  Interventions: Device: DEB+BMS
- POBA+DES (Active Comparator): conventional balloon predilation and drug-eluting stent implantation
  Interventions: Device: POBA+DES

INTERVENTIONS:
Device: DEB+BMS — drug-eluting balloon predilation and bare metal stent implantation
  Arms: DEB+BMS
Device: POBA+DES — conventional balloon predilation and drug-eluting stent implantation
  Arms: POBA+DES

SUMMARY:
The purpose of this study is to evaluate the efficacy of predilation with paclitaxel-eluting balloon and bare metal stent implantation VS conventional balloon and drug-eluting stent implantation in terms of restenosis

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* angina or stress test positive for ischemia
* de novo coronary stenosis>50%

Exclusion Criteria:

* recent myocardial infarction (<72h)
* severe chronic kidney disease
* allergy to Paclitaxel
* contraindication for combined antiplatelet treatment
* life expectancy <1 year
* hypersensitivity or contraindication to one of the study drugs
* lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
angiographic binary re-restenosis | 9 months
  incidence of angiographic binary re-restenosis

SECONDARY OUTCOMES:
Late luminal loss | 9 months
  incidence of late luminal loss assessed by angiography
major adverse cardiac events | 12 months
  incidence of major adverse cardiac events

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Bolognese, MD, Principal Investigator — San Donato Hospital
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy